CLINICAL TRIAL: NCT03019315
Title: The Analyses of Treatment Efficacy and Cost-effectiveness in Early-staged Ovarian Cancer Patients Treated With or Without Paclitaxel Regimens
Brief Title: The Analyses of Treatment Efficacy and Cost-effectiveness in Early-staged Ovarian Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201310006RIND
Record Dates: First submitted 2017-01-10; First posted 2017-01-12 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer; Chemotherapy; Response Rate; Survival
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

SUMMARY:
Adjuvant chemotherapy was introduced in patients with early-stage ovarian cancer. The benefit of standard chemotherapeutic regimens including taxane has not been established. This study was conducted to investigate the influences of regimens of front-line chemotherapy on on recurrence and survival for early-stage ovarian adenocarcinoma. Further, the study will analyze cost-effectiveness of different regimens

DETAILED DESCRIPTION:
Ovarian carcinoma has become more and more important in recent years because it is the leading cause of death among all gynecologic malignancies. The annual incidence rate of ovarian cancer in the United States was 11.8 per 100,000 and the death rate was 7.8 per 100,000 in 2009. According to the Department of Health Bureau's report, the incidence rate of ovarian cancer was 8.46 per 100,000 in 2010 and the death rate was 2.8 per 100,000. No specific symptoms, difficulty in early diagnosis, insufficient accurate tumor markers, and a lack of information regarding ovarian tumor biology all contribute to a poor prognosis.

The standard treatment for ovarian cancer is surgical tumor debulking, followed by platinum-containing chemotherapy. The conventional adjuvant chemotherapeutic regimens of ovarian cancer are platinum combined with cyclophosphamide. Whereas, platinum combined with paclitaxel has been identified to be a better adjuvant chemotherapeutic regimens for those advance-staged disease. In United States, platinum combined with paclitaxel has been used as standard adjuvant chemotherapeutic regimens for all of ovarian cancer patients for decades. However, many countries including Taiwan still use platinum combined with cyclophosphamide as adjuvant chemotherapeutic regimens for early-staged ovarian cancer patients. There is no comprehensive result to demonstrate the differences between these two regimens the fields of efficacy, side effects, survival, cost-effectiveness, and so on. So the investigators conduct this study to answer the questions. This study will firstly focus on the early-staged ovarian cancer patients to analyze the data from the National Health Insurance (NHI) databank. Further this study will then validate the results from NHI databank from the cancer registration system of National Taiwan University Hospital.

There are several aims in this proposal. First, the study will evaluate the differences of efficacy including the response rate, side effects, disease-free survival, and overall survival of the patients between these two chemotherapeutic regimens. Second, the cost-effectiveness of these two chemotherapeutic regimens will be identified. The results of this study will provide a more comprehensive picture of selecting optimal chemotherapeutic regimens for early-staged ovarian cancer patients. It can also be an important reference for the pay-off of National Health Insurance.

ELIGIBILITY:
Inclusion Criteria:

* (1) diagnosed at early stage, (2) treated with primary cytoreductive surgery followed by adjuvant platinum based chemotherapy

Exclusion Criteria:

* (1)patients with a history of cancer (2)patients had insufficient clinic-pathological and survival data regarding to disease prognosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ovarian cancer patients diagnosed between 1 January 1999 and 31 December 2020 without a history of cancer were identified from the catastrophic illness registry.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2015-01; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 5 years

SECONDARY OUTCOMES:
over all survival | 5 years
response rate | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Fang Cheng, Ph.D., Principal Investigator — Department of Obstetrics and Gynecology, College of Medicine, National Taiwan University, Taipei, Taiwan
Locations (1):
- National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No